CLINICAL TRIAL: NCT00193557
Title: Phase I Trial of Weekly Bortezomib (Velcade) in the Treatment of Patients With Refractory Multiple Myeloma
Brief Title: Weekly Bortezomib (Velcade) in the Treatment of Patients With Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI MM 06; 208538
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2009-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

INTERVENTIONS:
Drug: Bortezomib

SUMMARY:
This phase I study will evaluate the feasibility and toxicity of weekly bortezomib in the treatment of relapsed or refractory multiple Myeloma and determine whether a twice-weekly schedule of bortezomib is effective in producing responses in patients with stable disease or progression after weekly bortezomib

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be receive:

* Bortezomib

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Multiple Myeloma
* Received no more than 2 previous treatment regimens for multiple Myeloma
* ECOG performance status 0, 1, or 2
* Serum creatinine < 2.0mg/dL
* calculated or measured creatinine clearance > 30ml/minute
* Measurable or evaluable disease
* Provide written informed consent prior to receiving protocol therapy.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Moderate or severe peripheral neuropathy
* Other serious medical conditions
* Other active malignancies
* history of treatment for other invasive cancers
* Women who are pregnant or lactating

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-05; Primary Completion 2006-05 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
objective response rate

SECONDARY OUTCOMES:
progression-free survival
overall survival
Safety

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (2):
- United States (2):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Result] Hainsworth JD, Spigel DR, Barton J, Farley C, Schreeder M, Hon J, Greco FA. Weekly treatment with bortezomib for patients with recurrent or refractory multiple myeloma: a phase 2 trial of the Minnie Pearl Cancer Research Network. Cancer. 2008 Aug 15;113(4):765-71. doi: 10.1002/cncr.23606. PMID 18543319